CLINICAL TRIAL: NCT04050969
Title: Bariatric Atrial Restoration of Sinus Rhythm
Acronym: BAROS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult enrollment
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Paul Wang, Director, Stanford Electrophysiology and Arrhythmia Service, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID # 49225
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Atrial Fibrillation; Morbid Obesity
MeSH Terms: conditions — Atrial Fibrillation; Obesity, Morbid | interventions — Bariatric Surgery; Catheter Ablation

STUDY DESIGN:
Intervention Model Description: Patients will undergo screening and eligibility to make sure they meet all criteria for the trial. If patients meet all defined criteria, they will undergo informed consent and will be randomized with equal allocation to the catheter ablation only and bariatric surgery plus AF catheter ablation arms. Randomization will be stratified by site and type of AF (paroxysmal or persistent) using permuted blocks to limit effects of clinician variation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atrial Fibrillation (AF) Catheter Ablation-Group A (Active Comparator): Participants will undergo catheter ablation using either radiofrequency or cryo-ablation of pulmonary veins. Participants with persistent AF may also undergo roof and/or floor linear ablation with or without ablation of extra-pulmonary sites at the physician's discretion.
  Interventions: Procedure: Atrial Fibrillation (AF) Catheter Ablation
- Bariatric surgery prior to AF Catheter Ablation-Group B (Experimental): Participants will undergo either a Roux-en-Y gastric bypass or a laparoscopic sleeve gastrectomy. The choice of the procedure will be based on numerous factors including current practice, the surgeon's and participant's choice, BMI, and the presence of certain comorbidities and their severity such as GERD, kidney stones, and past surgical history. Participants will undergo standard preoperative evaluation including dietary consultation and psychological evaluation during the eligibility process.
  After bariatric surgery, in addition to routine post-surgical management, patients will follow up with cardiologist prior to AF catheter ablation.
  Interventions: Procedure: Bariatric surgery; Procedure: Atrial Fibrillation (AF) Catheter Ablation

INTERVENTIONS:
Procedure: Bariatric surgery — Participants will undergo either a laparoscopic sleeve gastrectomy or laparoscopic Roux-en-Y gastric bypass.
  Arms: Bariatric surgery prior to AF Catheter Ablation-Group B
Procedure: Atrial Fibrillation (AF) Catheter Ablation — Participants will undergo catheter ablation using either radiofrequency or cryoablation of pulmonary veins. Participants with persistent AF may also undergo roof and/or floor linear ablation with or without ablation of extrapulmonary sites at the physician's discretion.

SUMMARY:
The objective of this study is to determine whether bariatric surgery followed by Atrial Fibrillation (AF) catheter ablation is superior to AF catheter ablation alone in the management of atrial fibrillation in patients with morbid obesity.

DETAILED DESCRIPTION:
This will be a multicenter, randomized, controlled, 1:1 allocation trial comparing Atrial Fibrillation (AF) catheter ablation only (Group A) to those undergoing bariatric surgery six months prior to AF catheter ablation (Group B) in patients with paroxysmal or persistent AF who also have morbid obesity.

Participants will be followed for 12 months after their protocol-assigned catheter ablation. Scheduled visits Group A will be at baseline, 3, 6, and 12 months post AF ablation. Scheduled visits in Group B will be baseline, clinical visit prior AF ablation, and at 3, 6, and 12 months post AF ablation. At each post ablation visit the following data will be collected:

AT/AF recurrence determined by ambulatory monitoring, clinic visit, or hospitalization; Physical Exam (weight, height, vitals); 12 lead ECG; Medication Regimen; AF Symptom Severity Scale (AFSS); Quality of Life (AFEQT); Laboratory Testing; and Adverse Events

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic persistent or paroxysmal AF refractory to at least one antiarrhythmic agent
* EF > 40%
* BMI > 40 or BMI > 35 and at least one of the following co-morbidities:

  * Type 2 Diabetes Mellitus (by American Diabetes Association diagnostic criteria).
  * Systolic blood pressure of 130 mmHg and/or diastolic blood pressure 80 mmHg or higher despite medical treatment with maximal doses of three antihypertensive medications).
  * Refractory hyperlipidemia (acceptable levels of lipids unachievable with diet and maximum doses of lipid lowering medications).
  * Obesity-induced cardiomyopathy.
  * Clinically significant obstructive sleep apnea.
  * Obesity-related hypoventilation.
  * Pseudotumor cerebri (documented idiopathic intracerebral hypertension).
  * Severe arthropathy of spine and/or weight-bearing joints (when obesity prohibits appropriate surgical management of joint dysfunction treatable but for the obesity).
  * Hepatic steatosis without evidence of active inflammation.
  * Hypertriglyceridemia
  * Polycystic Ovary Syndrome (PCOS)
  * Asthma
  * Coronary Artery Disease (CAD)

Exclusion Criteria:

* Prior bariatric surgery
* Prior AF catheter ablation
* BMI > 65 kg/m2
* Contraindication to bariatric surgery or AF ablation
* Contraindication to therapeutic anticoagulation
* Sustained AF lasting more than 3 years
* Left atrial diameter of greater than or equal to 60 mm or LA volume greater than or equal to 60 ml/m2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Time to first recurrence of AF following a 3-month blanking period after the ablation. | Time to first recurrence of AF following a 3-month blanking period after the AF Catheter ablation.
  The primary outcome measure will be time to first recurrence of any atrial arrhythmia including AF, atrial flutter, or atrial tachycardia lasting longer than 30 seconds and occurring more than 3 months after AF ablation, without the use of antiarrhythmic medications. An episode of AF or atrial tachycardia will be considered part of the primary outcome analysis if it lasts longer than 30 seconds and is documented by any form of electrocardiographic monitoring, regardless of symptoms. A repeat catheter ablation procedure at any time will constitute a recurrence for the outcome analysis.

SECONDARY OUTCOMES:
Change in AF Burden off anti-arrhythmic agents monitor | Baseline (Initial), 3 months)
  The percentage of time in AF burden on the cardiac monitor will be calculated
Change in AF Burden off anti-arrhythmic agents monitor | Baseline (Initial), 6 months)
  The percentage of time in AF burden on the cardiac monitor will be calculated
Change in AF Burden off anti-arrhythmic agents monitor | Baseline (Initial), 12 months)
  The percentage of time in AF burden on the cardiac monitor will be calculated
Change from Baseline in AF Quality of Life Score | Baseline (Initial), 6 months
  Quality of Life will be assessed using a patient completed questionnaire, Cardiff Cardiac Ablation Patient Reported Outcome Measure (C-CAP) Questionnaire, pre-ablation (C-CAP1) and post ablation (C-CAP-2). The C-CAP score is a combined score of 16-18 items (0-30) with a higher score representing greater QOL.
Change from Baseline in AF Quality of Life Score | Baseline (Initial), 12 months
  Quality of Life will be assessed using a patient completed questionnaire, Cardiff Cardiac Ablation Patient Reported Outcome Measure (C-CAP) Questionnaire, pre-ablation (C-CAP1) and post ablation (C-CAP-2). The C-CAP score is a combined score of 16-18 items (0-30) with a higher score representing greater QOL.
Change from Baseline in AF symptom severity | Baseline (Initial), 6 months
  AF symptom burden will be assessed with the Atrial Fibrillation Symptoms Severity Scale. The AFSS is a patient self-reported questionnaire that contains 21 questions with 7 questions providing a calculated scores for AF symptom severity (0-35) with higher scores representing greater severity.
Change from Baseline in AF symptom severity | Baseline (Initial), 12 months
  AF symptom burden will be assessed with the Atrial Fibrillation Symptoms Severity Scale. The AFSS is a patient self-reported questionnaire that contains 21 questions with 7 questions providing a calculated scores for AF symptom severity (0-35) with higher scores representing greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Wang, MD, Principal Investigator — Director Stanford Electrophysiology and Arrhythmia Service, Stanford University; Dan E Azagury, MD, Principal Investigator — Assistant Professor of Surgery, Bariatric & Minimally Invasive Surgery
Locations (1):
- Stanford Health Care, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lavie CJ, Pandey A, Lau DH, Alpert MA, Sanders P. Obesity and Atrial Fibrillation Prevalence, Pathogenesis, and Prognosis: Effects of Weight Loss and Exercise. J Am Coll Cardiol. 2017 Oct 17;70(16):2022-2035. doi: 10.1016/j.jacc.2017.09.002. PMID 29025560
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- [Background] Abed HS, Wittert GA, Leong DP, Shirazi MG, Bahrami B, Middeldorp ME, Lorimer MF, Lau DH, Antic NA, Brooks AG, Abhayaratna WP, Kalman JM, Sanders P. Effect of weight reduction and cardiometabolic risk factor management on symptom burden and severity in patients with atrial fibrillation: a randomized clinical trial. JAMA. 2013 Nov 20;310(19):2050-60. doi: 10.1001/jama.2013.280521. PMID 24240932
- [Background] Middeldorp ME, Pathak RK, Meredith M, Mehta AB, Elliott AD, Mahajan R, Twomey D, Gallagher C, Hendriks JML, Linz D, McEvoy RD, Abhayaratna WP, Kalman JM, Lau DH, Sanders P. PREVEntion and regReSsive Effect of weight-loss and risk factor modification on Atrial Fibrillation: the REVERSE-AF study. Europace. 2018 Dec 1;20(12):1929-1935. doi: 10.1093/europace/euy117. PMID 29912366